CLINICAL TRIAL: NCT03440424
Title: An Open-Label, Parallel-Group Study to Evaluate the Pharmacokinetics of Lemborexant (E2006) and Its Metabolites in Subjects With Mild and Moderate Hepatic Impairment Compared to Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of Lemborexant (E2006) and Its Metabolites in Subjects With Mild and Moderate Hepatic Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-104
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2018-02

CONDITIONS: Hepatic Impairment
Keywords: mild hepatic impairment; moderate hepatic impairment; lemborexant; healthy participants; metabolites; E2006; pharmacokinetics
MeSH Terms: interventions — lemborexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Mild Hepatic Impairment (Child Pugh Class A) (Experimental): Participants with mild hepatic impairment will receive a single 10 milligram (mg) dose (1 × 10 mg lemborexant [E2006] tablet) in the morning with 240 milliliters (mL) of water following an overnight fast of at least 10 hours.
  Interventions: Drug: Lemborexant
- Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) (Experimental): Participants with moderate hepatic impairment will receive a single 10 mg dose (1 × 10 mg lemborexant [E2006] tablet) in the morning with 240 mL of water following an overnight fast of at least 10 hours.
  Interventions: Drug: Lemborexant
- Cohort C: Healthy Participants (Control) (Experimental): Healthy participants matched to participants with hepatic impairment in Cohorts A and B (matched with regards to age, sex, body mass index [BMI]) will receive a single 10 mg dose (1 × 10 mg lemborexant [E2006] tablet) in the morning with 240 mL of water following an overnight fast of at least 10 hours.
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — oral tablet

SUMMARY:
This study will be conducted to assess the effect of mild and moderate hepatic impairment on the pharmacokinetics (PK) of lemborexant after a single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Participants:

* Male or female participants, ages 18 to 79, inclusive, at the time of informed consent
* Body Mass Index (BMI) between 18 and 40 kilograms per meters squared, inclusive, at Screening
* Voluntary agreement to provide written informed consent, and the willingness and ability to comply with all aspects of the protocol
* Nonsmokers or smokers who smoke 20 cigarettes or less per day
* For Cohorts A and B: stable (without any change in disease status for at least 60 days prior to study Screening) hepatic impairment conforming to Child-Pugh classification A or B, respectively, and documented by medical history and a physical examination
* For Cohort C: healthy participants matched to participants with hepatic impairment with regard to age (±10 years), sex, and BMI (±20%), and as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECG), and clinical laboratory determinations

Exclusion Criteria:

Exclusion Criteria for All Participants:

* Females who are breastfeeding or pregnant at Screening or Baseline
* Females of childbearing potential who did not use a highly effective method of contraception within 28 days before study entry, or who did not agree to use an approved method of contraception from 28 days before study entry, throughout the entire study period, and for 28 days after study drug discontinuation. Approved (highly effective) methods of contraception for this study included at least one of the following: 1. Total abstinence (if it was their preferred and usual lifestyle); 2. An intrauterine device or intrauterine hormone-releasing system (IUS); 3. A double-barrier method of contraception such as condom plus diaphragm with spermicide; 4. A contraceptive implant; 5. An oral contraceptive (with additional barrier method). Participant must have been on a stable dose of the same oral contraceptive product for at least 28 days before dosing, throughout the study, and for 28 days after study drug discontinuation; 6. Have a vasectomized partner with confirmed azoospermia. (Note: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* Known to be positive for human immunodeficiency virus
* Currently enrolled in another clinical study or used any investigational drug or device within 4 weeks, or 5 times the half-life of the investigational drug (whichever is longer), preceding informed consent
* Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing until study discharge
* Intake of herbal preparations containing St. John's Wort within 4 weeks prior to dosing until study discharge
* Intake of nutritional supplements (including herbal preparations), foods or beverages that may affect cytochrome P3A enzyme (e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 1 week before dosing until study discharge
* Intake of beverages, food, or other products that contain caffeine from 24 hours before until 48 hours after dosing with lemborexant
* Engagement in strenuous exercise (e.g., moving large bulky items, bodybuilding) within 2 weeks prior to check-in until study discharge
* History of clinically significant drug or food allergies, or is presently experiencing significant seasonal allergies
* A prolonged QT/corrected QT (QTc) interval (QTc >480 milliseconds) demonstrated on ECG at Screening or Baseline (Day -1)
* Any major surgery within 4 weeks of study drug administration
* Any history of abdominal surgery that may affect pharmacokinetics of lemborexant (e.g., hepatectomy, nephrectomy, digestive organ resection)
* Inability to tolerate oral medication
* Inability to tolerate venous access and/or venipuncture
* Unwilling to abide by the study requirements, or in the opinion of the investigator, is not likely to complete the study

Additional Exclusion Criteria for Hepatically Impaired Participants (Cohorts A and B):

In addition to the Exclusion Criteria listed above for all participants, other standard exclusion criteria for participants with hepatic impairment will be used. These include:

* Any significant acute medical illness (such as new conditions or exacerbation of pre-existing conditions) within 8 weeks of dosing
* Medical conditions which are not adequately and stably controlled on stable doses of medications or which, in the clinical opinion of the Principal Investigator, may interfere with study procedures or participant safety within 4 weeks before dosing (e.g., psychiatric disorders and disorders of the gastrointestinal tract, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism)
* History of esophageal and gastric variceal bleeding within the past 6 months unless the participant has completed a course of endoscopic therapy with the appropriate documentation (e.g., endoscopy report) of successful ablation of esophageal varices; participants with esophageal varices may be included if not bleeding within the past 6 months or have been treated adequately by ablation therapy, as specified above.
* Spontaneous bacterial peritonitis within 3 months of dosing
* Treatment with plasmapheresis within 6 months of dosing
* Primarily cholestatic liver diseases (e.g., primary biliary cirrhosis or primary sclerosing cholangitis)
* Current or recent (within 3 months prior to Screening) history of significant gastrointestinal disease other than that secondary to hepatic impairment
* Autoimmune liver disease
* Active alcoholic hepatitis determined either clinically or by histology
* History of hepatoma or metastatic disease of the liver
* Presence of severe ascites or edema
* Presence of hepatopulmonary syndrome or hydrothorax, or hepatorenal syndrome
* Known significant bleeding diathesis that could preclude multiple venipunctures (international normalization ratio >2.5)
* Creatinine clearance <60 milliliters per minute at Screening or Baseline as calculated using Cockroft and Gault Equation
* The participant's standard therapy/concomitant medication for diseases related to cirrhosis has not remained stable/unchanged for at least 14 days before the first dose of study drug
* History of drug or alcohol dependency or abuse within 4 weeks prior to Screening, or those who have a positive urine drug test or breath alcohol test at Screening or Baseline unless a prescribed medication for the underlying condition is the cause of the positive urine screen

Additional Exclusion Criteria for Healthy Participants (Cohort C):

In addition to the Exclusion Criteria listed above for all participants, other standard exclusion criteria for healthy participants in Phase 1 studies will be used. These include:

* Presence of active liver disease, or acute liver injury, as indicated by (1) an abnormal liver function test, or (2) clinical or laboratory signs of active viral hepatitis (including B and C, as demonstrated by positive serology at Screening)
* Clinically significant illness, within 4 weeks prior to dosing, that requires medical treatment or may influence the outcome of the study; e.g., psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
* Any abnormal finding based on physical examination, assessment of vital signs, ECG, or laboratory test results that require treatment or clinical follow-up based on the investigator's opinion
* History of drug or alcohol use disorder within the 2 years prior to Screening, or those who have a positive urine drug test or breathalyzer alcohol test at Screening or Baseline
* Use of any prescription drugs within 4 weeks prior to dosing until study discharge
* Intake of any over-the-counter medications within 2 weeks prior to dosing until study discharge

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 26 January 2018 to 23 April 2018.
Pre-assignment Details: A total of 28 participants were screened, of which 4 were screen failures, and 24 were enrolled and received the study treatment.
Groups:
- Cohort A: Mild Hepatic Impairment (Child Pugh Class A): Participants with mild hepatic impairment (Child-Pugh Class A, score 5 to 6) received lemborexant 10 milligrams (mg) administered as a tablet, orally in the morning on Day 1 of the 14-day Treatment Period. The Child-Pugh Score is a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon albumin, ascites, total bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
- Cohort B: Moderate Hepatic Impairment (Child Pugh Class B): Participants with moderate hepatic impairment (Child-Pugh Class B, score 7 to 9) received lemborexant 10 mg administered as a tablet, orally in the morning on Day 1 of the 14-day Treatment Period. The Child-Pugh Score is a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon albumin, ascites, total bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
- Cohort C: Healthy Participants (Control): Healthy participants matched to participants with hepatic impairment in Cohorts A and B (with regards to age, sex, body mass index [BMI]) received lemborexant 10 mg administered as a tablet, orally in the morning on Day 1 of the 14-day Treatment Period.
Period: Overall Study
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was the group of participants who were dosed with the test drug and had atleast 1 postdose safety assessment.
Groups:
- Cohort A: Mild Hepatic Impairment (Child Pugh Class A): Participants with mild hepatic impairment (Child-Pugh Class A, score 5 to 6) received lemborexant 10 mg administered as a tablet, orally in the morning on Day 1 of the 14-day Treatment Period. The Child-Pugh Score is a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon albumin, ascites, total bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
- Cohort C: Healthy Participants (Control): Healthy participants matched to participants with hepatic impairment in Cohorts A and B (with regards to age, sex, BMI) received lemborexant 10 mg administered as a tablet, orally in the morning on Day 1 of the 14-day Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (10.5) | 61.4 (5.7) | 56.8 (8.3) | 58.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 6 | 6 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 5 | 12
  Not Hispanic or Latino | 3 | 6 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Plasma Concentration of Lemborexant
Description: Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. Plasma pharmacokinetic (PK) data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: The PK Analysis Set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter (ng/mL) | 62.9 (34.9) | 48.7 (37.7) | 39.8 (31.1)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 157.86, 90% CI 2-sided [118.18 to 210.87] — Percent ratio of geometric mean was calculated by dividing the geometric mean of test by geometric mean of reference, then multiplying the value by 100
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 122.20, 90% CI 2-sided [91.49 to 163.24] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: AUC(0-8 Hours): Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours Postdose of Lemoborexant
Description: Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-8 hours) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
hour nanogram per milliliter (h*ng/mL) | 163 (32.8) | 138 (13.8) | 133 (25.1)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 122.31, 90% CI 2-sided [98.95 to 151.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 103.24, 90% CI 2-sided [83.53 to 127.61] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC(0-72 Hours): Area Under the Plasma Concentration-Time Curve From Time Zero to 72 Hours Postdose of Lemoborexant
Description: Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-72 hours) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 383 (46.1) | 352 (13.0) | 306 (25.0)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 125.26, 90% CI 2-sided [96.76 to 162.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 115.20, 90% CI 2-sided [88.98 to 149.13] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: AUC(0-t Hours): Area Under Plasma Concentration Versus Time Curve From Time Zero to Time of Last Quantifiable Concentration of Lemborexant
Description: Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-t hours) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 574 (50.7) | 651 (25.6) | 435 (33.2)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 131.91, 90% CI 2-sided [96.46 to 180.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 149.52, 90% CI 2-sided [109.34 to 204.47] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC(0-inf): Area Under Plasma Concentration Versus Time Curve From Time Zero to Infinity of Lemborexant
Description: Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-inf) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: The PK Analysis Set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least 1 PK parameter. Here "Overall number of participants analyzed" signifies the participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 7 | 6 | 8
h*ng/mL | 567 (52.0) | 696 (34.6) | 453 (33.9)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 125.03, 90% CI 2-sided [87.96 to 177.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 153.56, 90% CI 2-sided [106.39 to 221.66] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUCu: AUC(0-inf) Values Adjusted by Unbound Fraction in Plasma of Lemborexant
Description: AUCu was defined as the AUC(0-inf) adjusted by unbound fraction in plasma, and calculated by multiplying the value of AUC(0-inf) with plasma protein unbound fraction (fu). Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUCu was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 7 | 6 | 8
h*ng/mL | 34.9 (52.6) | 45.1 (42.6) | 27.1 (36.8)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 128.88, 90% CI 2-sided [88.35 to 188.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); Test type: Other; Percent ratio of geometric mean = 166.55, 90% CI 2-sided [112.31 to 246.99] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Cmax: Maximum Plasma Concentration of Lemborexant's Metabolites M4, M9, and M10
Description: Blood samples were analyzed for the amount of lemborexant's metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  M4 | 7.73 (36.4) | 5.74 (46.7) | 7.97 (33.0)
  M9 | 4.49 (45.1) | 3.50 (46.4) | 5.33 (28.9)
  M10 | 3.52 (44.4) | 2.84 (38.4) | 3.71 (34.8)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 96.97, 90% CI 2-sided [70.15 to 134.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 72.05, 90% CI 2-sided [52.12 to 99.60] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 84.36, 90% CI 2-sided [60.21 to 118.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 65.70, 90% CI 2-sided [46.89 to 92.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 94.74, 90% CI 2-sided [68.37 to 131.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 76.56, 90% CI 2-sided [55.24 to 106.09] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration of Lemborexant and Its Metabolites M4, M9, M10
Description: Blood samples were analyzed for the amount of lemborexant and its metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
hours
  Lemborexant | 1.00 [0.50 to 1.50] | 1.00 [0.50 to 3.00] | 1.25 [0.50 to 4.00]
  M4 | 1.75 [1.00 to 4.00] | 1.75 [1.00 to 4.00] | 2.00 [1.00 to 4.00]
  M9 | 1.25 [1.00 to 3.00] | 1.25 [1.00 to 4.00] | 1.50 [1.00 to 4.00]
  M10 | 4.00 [2.00 to 24.00] | 3.00 [1.00 to 4.00] | 4.00 [4.00 to 24.00]

9. Secondary Outcome: AUC(0-8 Hours): Area Under Plasma Concentration Versus Time Curve From Time Zero to 8 Hours Postdose of Lemborexant's Metabolites M4, M9, and M10
Description: Blood samples were analyzed for the amount of lemborexant's metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-8 hours) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL
  M4 | 44.2 (27.2) | 31.0 (34.4) | 44.6 (28.6)
  M9 | 17.5 (29.2) | 14.0 (31.1) | 22.2 (19.3)
  M10 | 21.4 (40.7) | 16.3 (35.1) | 22.6 (40.4)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 99.14, 90% CI 2-sided [76.91 to 127.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 69.66, 90% CI 2-sided [54.03 to 89.79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 78.98, 90% CI 2-sided [62.88 to 99.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 63.20, 90% CI 2-sided [50.31 to 79.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 94.56, 90% CI 2-sided [68.50 to 130.51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 71.81, 90% CI 2-sided [52.03 to 99.12] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: AUC(0-72 Hours): Area Under Plasma Concentration Versus Time Curve From Time Zero to 72 Hours Postdose of Lemborexant's Metabolites M4, M9, and M10
Description: Blood samples were analyzed for the amount of lemborexant's metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-72 hours) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL
  M4 | 153 (36.7) | 123 (19.5) | 144 (26.8)
  M9 | 52.1 (29.1) | 52.5 (18.9) | 69.1 (18.0)
  M10 | 167 (41.3) | 130 (23.0) | 175 (35.3)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 106.70, 90% CI 2-sided [83.95 to 135.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 85.68, 90% CI 2-sided [67.41 to 108.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 75.41, 90% CI 2-sided [62.28 to 91.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 76.00, 90% CI 2-sided [62.76 to 92.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 95.55, 90% CI 2-sided [71.92 to 126.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 74.48, 90% CI 2-sided [56.06 to 98.94] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: AUC(0-t Hours): Area Under Plasma Concentration Versus Time Curve From Time Zero to t Hours Postdose of Lemborexant's Metabolites M4, M9, and M10
Description: Blood samples were analyzed for the amount of lemborexant's metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-t hours) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL
  M4 | 208 (45.8) | 191 (20.6) | 184 (31.3)
  M9 | 69.7 (34.9) | 89.6 (23.0) | 88.7 (21.4)
  M10 | 334 (42.8) | 321 (19.9) | 305 (41.5)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 113.04, 90% CI 2-sided [85.16 to 150.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 103.74, 90% CI 2-sided [78.16 to 137.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 78.62, 90% CI 2-sided [62.57 to 98.78] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 101.00, 90% CI 2-sided [80.38 to 126.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 109.49, 90% CI 2-sided [81.07 to 147.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 105.20, 90% CI 2-sided [77.89 to 142.08] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: AUC(0-inf): Area Under Plasma Concentration Versus Time Curve From Time Zero to Inf Hours Postdose of Lemborexant's Metabolites M4, M9, and M10
Description: Blood samples were analyzed for the amount of lemborexant's metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. AUC(0-inf) was calculated by the linear-up log-down trapezoidal method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: The PK Analysis Set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least 1 PK parameter. Here "Number analyzed" signifies participants who were evaluable for this outcome measure for different metabolites M4, M9, and M10.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL
  M4: number analyzed (Participants) | 6 | 6 | 8
  M4 | 220 (50.3) | 223 (21.3) | 191 (31.6)
  M9: number analyzed (Participants) | 7 | 6 | 7
  M9 | 72.6 (34.7) | 108 (21.6) | 92.5 (23.5)
  M10: number analyzed (Participants) | 6 | 5 | 8
  M10 | 304 (27.7) | 332 (17.9) | 320 (41.9)
Statistical Analysis 1: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 115.38, 90% CI 2-sided [83.51 to 159.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M4 metabolite; Test type: Other; Percent ratio of geometric mean = 116.97, 90% CI 2-sided [84.66 to 161.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 78.46, 90% CI 2-sided [61.06 to 100.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M9 metabolite; Test type: Other; Percent ratio of geometric mean = 116.76, 90% CI 2-sided [89.95 to 151.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Mild Hepatic Impairment (Child Pugh Class A) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 94.97, 90% CI 2-sided [70.31 to 128.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) vs Cohort C: Healthy Participants (Control); M10 metabolite; Test type: Other; Percent ratio of geometric mean = 103.59, 90% CI 2-sided [75.43 to 142.28] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: T1/2: Terminal Plasma Phase Half-life of Lemborexant and Its Metabolites M4, M9, M10
Description: Terminal plasma half-life is the time required for plasma/blood concentration to decrease by 50%. This is not the time required to eliminate half the administered dose. Blood samples were analyzed for the amount of lemborexant and its metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: The PK Analysis Set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least 1 PK parameter. Here "Number analyzed" signifies participants who were evaluable for this outcome measure for lemborexant and its metabolites (M4, M9, and M10).
Measure: Median (Full Range); unit: hrs
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
hrs
  Lemborexant: number analyzed (Participants) | 7 | 6 | 8
  Lemborexant | 92.7 [33.4 to 104] | 115 [72.8 to 144] | 71.1 [40.4 to 88.9]
  M4: number analyzed (Participants) | 6 | 6 | 8
  M4 | 69.2 [26.7 to 95.1] | 102 [75.6 to 112] | 68.1 [16.7 to 95.3]
  M9: number analyzed (Participants) | 7 | 6 | 7
  M9 | 49.0 [26.4 to 102] | 88.4 [70.0 to 126] | 49.7 [14.0 to 72.7]
  M10: number analyzed (Participants) | 6 | 5 | 8
  M10 | 71.0 [40.3 to 88.9] | 96.8 [67.4 to 118] | 69.3 [32.3 to 90.7]

14. Secondary Outcome: CL/F: Apparent Total Body Clearance of Lemborexant
Description: CL/F is the clearance for parent lemborexant only and was calculated as Dose/[AUC 0-inf]. Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: The PK Analysis Set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least 1 PK parameter. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 7 | 6 | 8
Liter per hour (L/hr) | 17.6 (52.0) | 14.4 (34.6) | 22.1 (33.9)

15. Secondary Outcome: Vz/F: Apparent Volume of Distribution of Lemborexant
Description: The apparent volume of distribution gives information about amount of lemborexant distributed in body tissue rather than the blood/plasma. Vz/F for parent lemborexant only was calculated as Dose/(AUC0-inf multiplied by elimination rate constant[λz]). Area under the plasma concentration-time curve from time zero to infinity, calculated(AUC0-inf) as AUC0-t + AUCextra. AUCextra represents an extrapolated value obtained by Clast/λz, where Clast: plasma concentration at last sampling time point at which measured plasma concentration is at or above LLQ. λz is the elimination rate constant. Elimination rate constant obtained from linear regression of terminal phase of log transformed concentration-time data. A minimum of three points is required to calculate λz. Blood samples were analyzed for amount of lemborexant in plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 7 | 6 | 8
Liter (L) | 1880 (72.7) | 2170 (13.5) | 2130 (30.1)

16. Secondary Outcome: MPR: Metabolite-to-Parent Ratios of AUC(0-inf) for Lemborexant's Metabolites M4, M9, and M10
Description: The MPR is the ratio of AUC(0-inf) of the individual lemborexant metabolites (M4, M9, M10) to AUC(0-inf) of lemborexant, corrected for molecular weights. Blood samples were analyzed for the amount of lemborexant metabolites in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: The PK Analysis Set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least 1 PK parameter. Here "Number analyzed" signifies participants who were evaluable for the outcome measure for each metabolite (M4, M9, and M10).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
ratio
  M4: number analyzed (Participants) | 6 | 5 | 8
  M4 | 0.343 (2.90) | 0.289 (23.4) | 0.405 (11.5)
  M9: number analyzed (Participants) | 7 | 5 | 7
  M9 | 0.123 (19.0) | 0.144 (17.4) | 0.198 (22.0)
  M10: number analyzed (Participants) | 6 | 5 | 8
  M10 | 0.600 (15.3) | 0.502 (20.4) | 0.680 (18.9)

17. Secondary Outcome: fu: Plasma Protein Unbound Fraction of Lemborexant and Its Metabolites M4, M9, and M10
Description: Unbound fraction of drug in plasma was calculated as 100 percent (%) - mean percent of lemborexant and its metabolites M4, M9, and M10 bound to plasma protein for each participant. Blood samples were analyzed for the amount of lemborexant and its metabolites (M4, M9, M10) in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % (percent) unbound
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 8 | 8 | 8
% (percent) unbound
  Lemborexant | 0.0630 (14.2) | 0.0650 (11.4) | 0.0597 (15.3)
  M4 | 0.247 (7.77) | 0.247 (12.4) | 0.230 (12.8)
  M9 | 0.146 (14.0) | 0.142 (9.61) | 0.136 (15.8)
  M10 | 0.0765 (15.4) | 0.0754 (16.6) | 0.0669 (20.2)

18. Secondary Outcome: CLu/F: Apparent Clearance Relative to the Unbound Plasma Concentration Based on AUCu of Lemborexant
Description: Unbound fraction of drug in plasma was calculated as 100% - mean percent of lemborexant bound to plasma protein for each participant. Blood samples were analyzed for the amount of lemborexant in the plasma. Plasma concentration-time data were measured by validated LC-MS/MS method. Plasma PK data were analyzed using a non-compartmental method of analysis.
Time Frame: Day 1: Predose, 0.5 up to 312 hours postdose
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
Number analyzed (Participants) | 7 | 6 | 8
L/h | 287 (52.6) | 222 (42.6) | 370 (36.8)

ADVERSE EVENTS:
Time Frame: From the date of first dose up to 28 days after the last dose of study drug (up to 42 days)
Arm/Group | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) | Cohort C: Healthy Participants (Control)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 6/8 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Mild Hepatic Impairment (Child Pugh Class A) (N=8) | Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) (N=8) | Cohort C: Healthy Participants (Control) (N=8)
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 7 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03440424/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT03440424/SAP_003.pdf